CLINICAL TRIAL: NCT00820456
Title: Angle Interleaved Projection Reconstruction With K-Space Weighted Image Reconstruction for Dynamic Contrast MRI of Cancer Therapy Response
Brief Title: Metastatic Colorectal Cancer: Treatment Response With Dynamic Contrast MRI
Status: Terminated | Type: Observational
Why Stopped: Study did not meet enrollment goals.
Sponsor: American College of Radiology (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: ACRIN PA 4002; SAP #4100031303
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Neoplasm; Hepatic Neoplasm
Keywords: colorectal cancer; colorectal neoplasm; colorectal neoplasms; metastasis; metastases; liver; hepatic metastasis; liver metastasis; perfusion imaging; MRI; magnetic resonance imaging; dynamic contrast enhanced MRI; dynamic contrast enhanced magnetic resonance imaging
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Colorectal Cancer, Hepatic Metastasis: Eligible participants in Arm A enrolled in this imaging study will: be older than 18, have metastatic colorectal cancer with at least one hepatic lesion, and be treated with FOLFOX in combination with bevacizumab.
  Interventions: Other: DCE-MRI
- Primary Tumor Undefined, Hepatic Metastasis: Eligible participants in Arm B enrolled in this imaging study will: be older than 18, must have prior histological documentation of any types of cancer with metastasis to the liver, and must be in stable treatment conditions prior to and between scans.
  Interventions: Other: DCE-MRI

INTERVENTIONS:
Other: DCE-MRI — Participants will receive two (2) dynamic contrast enhanced magnetic resonance imaging (DCE-MRI) prior to chemotherapy and one (1) DCE-MRI after the first cycle of chemotherapy. Participants will be followed for up to 2 years after the initiation of chemotherapy or until disease progression.
  Other Names: Dynamic Contrast Enhanced Magnetic Resonance Imaging; dynamic contrast MRI; perfusion MRI; perfusion imaging

SUMMARY:
The objectives for this study include:

* Testing a unique way of imaging people with colorectal cancer and other cancers that has spread to the liver using magnetic resonance imaging (MRI);
* Seeing if the MRI process can be used across multiple imaging platforms;
* Determining whether the results of the imaging can be reproduced;
* Reviewing how MRI results relate to cancer response to combination therapy and to clinical endpoints.

DETAILED DESCRIPTION:
This study will investigate the use of projection reconstruction dynamic contrast-enhanced MRI (DCE-MRI) as a surrogate marker of tumor vascularity in patients treated with the antiangiogenic agent bevacizumab. DCE-MRI is gaining popularity as a method to assess the functional response of tumors to agents targeting the vascular endothelial growth factor (VGEF) pathways. DCE-MRI measurements have been proposed as a non-invasive measure of both tumor biologic activity and (in the case of antivascular therapy) early response to treatment. A number of phase I and II studies demonstrate the ability for DCE-MRI to detect perfusion changes associated with tumor biologic response to vascularly targeted agents. It has been suggested that pre-treatment DCE-MRI might identify tumors with high intrinsic perfusion and that these tumors will be more likely to respond to antivascular-based therapies. However, the current use of DCE-MRI in clinical settings is challenging. Trade-offs between spatial coverage, time, and spatial resolution make this technique difficult to implement in human studies and may limit its reliability. The use of projection reconstruction-based acquisition can mitigate the need for these trade-offs and can simultaneously provide high temporal and spatial resolution data for DCE-MRI analysis.

ELIGIBILITY:
Arm A: Inclusion Criteria:

* Participants must be >18 years old;
* Participants must have an ECOG performance status of 0-1;
* Participants must not be pregnant or breastfeeding;
* Participants must have prior histological documentation of adenocarcinoma of the colon or rectum;
* Participants must be commencing chemotherapy with FOLFOX plus bevacizumab;
* Participants must not have had prior exposure to bevacizumab. Prior systemic chemotherapy with other agents is allowed. The last dose of systemic chemotherapy must have been > 3 months prior to study entry;
* Participants with prior radiotherapy or other prior local therapy to the liver (radioablation therapy, chemoembolic therapy) are acceptable. They must be at least 4 weeks past the last administration of such therapy;
* Participants must be at least 4 weeks past any major surgery, including surgery to the liver;
* Participants with prior malignancies other than colon cancer are allowed, provided they have been treated with curative intent, and have no evidence of recurrence of that malignancy;
* Participants must have a life expectancy of greater than 3 months;
* Participants must have the ability to understand and the willingness to sign a written informed consent form.

Arm B: Inclusion Criteria

* Participants must be >18 years old;
* Participants must have an ECOG performance status of 0-1;
* Participants must not be pregnant or breastfeeding;
* Participants must have prior histological documentation of any types of cancer with metastasis to the liver (see Imaging Criteria below);
* Participants must be projected to be within a stable treatment condition prior to and between scans (see section 4.3 for definition of stable treatment condition);
* Participants must be at least 4 weeks past any major surgery, including surgery to the liver;
* Participants must have a life expectancy of greater than 3 months;
* Participants must have the ability to understand and the willingness to sign a written informed consent form.

Imaging Criteria:

* Participants must have at least one hepatic lesion greater than or equal to 3 cm in maximal diameter on cross sectional imaging study (CT or MRI) performed within 4 weeks prior to study enrollment;
* Participants must have at least one qualifying liver lesion (i.e. one greater than or equal to 3 cm) that has been confirmed metastatic adenocarcinoma of the colon or rectum based on one of the following criteria:

  * Histologic (FNA or core biopsy) proof of malignancy compatible with metastasis from a colorectal carcinoma; OR
  * Demonstration of imaging features of tumor metastasis to the liver, including at least one of the following:

    1. evidence of heterogeneous enhancement or central tumor necrosis by CT or MRI;
    2. previously demonstrated interval enlargement of the lesion by >25% in the longest diameter;
    3. PET image demonstrating metabolic activity characteristic of malignancy (FDG uptake greater than that of background liver).
* For participants who have undergone local hepatic surgical, radiation, ablative, or embolic therapy, the date of qualifying imaging study(ies) or qualifying biopsy must be at least 30 days after the last instance of such local therapy. Furthermore, cross-sectional imaging performed at least 30 days after such local therapy must demonstrate an area of residual viable tumor (as judged by enhancing tissue following contrast administration) with longest diameter ≥ 3cm in at least one cross-sectional axis.

Arms A and B (Unless Otherwise Indicated): Exclusion Criteria:

* Patients with contraindication to MRI, including:

  1. Contraindicated metallic device, including pacemaker, non-MRI compatible aneurysm clip, other non-MRI compatible mechanical and/or electrical device, or metallic fragments;
  2. Patients with severe claustrophobia (patients with milder forms of claustrophobia that can be successfully allayed with oral anxiolytic therapy are allowed);
* Patients with contraindication to gadolinium, including:

  a) Hypersensitivity to gadolinium-containing MR contrast agents;
* Severe impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73 m2 and/or on dialysis;
* Patients with severely compromised pulmonary, cardiovascular, or mental status. Patients must not have severe congestive heart failure (defined as New York Heart Association Class II or greater);
* For Arm A only: Any other major medical illness that, in the investigator's opinion, would: (1) prevent administration or completion of institution's standard of care FOLFOX/bevacizumab therapy; (2) prevent administration or completion of protocol-specified imaging; and/or (3) interfere with follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At each participating site, at least one oncologist treating patients with adenocarcinoma of the colon and rectum must agree to serve as a co-investigator on the study. However, all oncologists directly or indirectly affiliated with the participating institution may serve as a source of participants for this trial. Patients with adenocarcinoma of the colon or rectum metastatic to the liver who are present candidates for FOLFOX plus bevacizumab are eligible to enroll in this imaging trial in Arm A. Patients with any primary carcinoma with metastatic disease to the liver who are in stable treatment condition prior to and between scnas are eligible to enroll in this imaging trial in Arm B.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2009-12-31 (Actual); Study Completion 2009-12-31 (Actual)

PRIMARY OUTCOMES:
To determine the reproducibility of DCE-MRI measures of tumor Ktrans, kep, and ve for colorectal metastases to the liver (Arm A) and any cancer metastatic to the liver (Arm B), using projection interleaved back-projection DCE-MRI techniques. | Three (3) DCE-MRI scans (two separate pre-treatment and one post-treatment DCE-MRI exams [post-treatment defined as after the first cycle of chemotherapy with bevacizumab])
To determine the alteration in tumor vascularity (assessed by percentage change in tumor Ktrans) in Arm A participants with metastatic colorectal cancer to the liver after one cycle of chemotherapy including bevacizumab compared to baseline Ktrans value. | Two (2) DCE-MRI scans (baseline pre-treatment and post-treatment DCE-MRI exams [post-treatment defined as after the first cycle of chemotherapy with bevacizumab])

SECONDARY OUTCOMES:
To determine the relationship between initial tumor vascularity (absolute tumor Ktrans) and change in tumor vascularity (percentage change in tumor Ktrans after one cycle of chemotherapy) and PFS in participants in Arm A. | Two (2) DCE-MRI scans (baseline pre-treatment and post-treatment DCE-MRI exams [post-treatment defined as after the first cycle of chemotherapy with bevacizumab]) with follow-up
To evaluate the perfusional difference between the dominant tumor and the global tumor burden (Arms A and B). | Three (3) DCE-MRI scans (two separate pre-treatment and one post-treatment DCE-MRI exams [post-treatment defined as after the first cycle of chemotherapy with bevacizumab])
To evaluate the feasibility of exporting back-projection DCE-MRI imaging across multiple MRI scanner vendor platforms for use in a multi-site chemotherapy trial. | Three (3) DCE-MRI scans (two separate pre-treatment and one post-treatment DCE-MRI exams [post-treatment defined as after the first cycle of chemotherapy with bevacizumab])
To determine the functional status as a predictor of response or disease-free survival in participants in Arm A. | Three (3) DCE-MRI scans (two separate pre-treatment and one post-treatment DCE-MRI exams [post-treatment defined as after the first cycle of chemotherapy with bevacizumab]) with follow-up for response and disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rosen, MD, PhD, Principal Investigator — University of Pennsylvania; Larry Dougherty, PhD, Study Chair — University of Pennsylvania; Donald Mitchell, MD, Study Chair — Thomas Jefferson University; Peter J O'Dwyer, MD, Study Chair — University of Pennsylvania; Michael D Feldman, MD, PhD, Study Chair — University of Pennsylvania
Locations (5):
- United States (5):
  - Penn State University Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania